CLINICAL TRIAL: NCT04573751
Title: Intracoronary Administration of Epinephrine and Verapamil in the Refractory No-reflow Phenomenon in Patients With Acute Myocardial Infarction: The EPIVER Randomized Controlled Trial
Brief Title: The EPIVER Randomized Controlled Trial
Acronym: EPIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIVER
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: ST Elevation Myocardial Infarction; Percutaneous Coronary Intervention; No-Reflow Phenomenon
Keywords: Primary PCI; No-reflow; Intracoronary epinephrine
MeSH Terms: conditions — ST Elevation Myocardial Infarction; No-Reflow Phenomenon | interventions — Standard of Care; Epinephrine; Verapamil; Evoked Potentials, Visual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard therapy (Sham Comparator): No intracoronary epinephrine and verapamil
  Interventions: Drug: Standard therapy
- Epinephrine (Active Comparator): Intracoronary bolus epinephrine injection requires two ampoules each of 1:1,000 epinephrine (1 μg/mL) diluted into 100 mL of normal saline solution (to 20 μg/mL epinephrine solution); therefore, a 5-mL syringe contains 100 μg of epinephrine. Intracoronary epinephrine will be administered at a dose of 100 μg and at a lower dose of 80 μg in patients with blood pressure >160 mmHg
  Interventions: Drug: Epinephrine
- Verapamil (Active Comparator): Intracoronary verapamil is administered at a dose of 0.5 mg.
  Interventions: Drug: Verapamil
- Epinephrine + verapamil (Active Comparator): Intracoronary administration of epinephrine at a dose of 80-100 μg and verapamil at a dose of 0.5 mg.
  Interventions: Drug: Epinephrine + verapamil

INTERVENTIONS:
Drug: Standard therapy — Standard therapy as follows: adenosine, nitroglycerine, thrombus aspiration/extraction, and platelet IIb/IIIa receptor inhibitors.
  Other Names: Control
  Arms: Standard therapy
Drug: Epinephrine — Standard therapy plus epinephrine as follows: epinephrine, adenosine, nitroglycerine, thrombus aspiration/extraction, and platelet IIb/IIIa receptor inhibitors.
  Other Names: Epi
  Arms: Epinephrine
Drug: Verapamil — Standard therapy plus verapamil as follows: verapamil, adenosine, nitroglycerine, thrombus aspiration/extraction, and platelet IIb/IIIa receptor inhibitors.
  Other Names: Ver
  Arms: Verapamil
Drug: Epinephrine + verapamil — Standard therapy plus epinephrine + verapamil as follows: epinephrine, verapamil, adenosine, nitroglycerine, thrombus aspiration/extraction, and platelet IIb/IIIa receptor inhibitors.
  Other Names: Epi+Ver
  Arms: Epinephrine + verapamil

SUMMARY:
The trial aims to estimate the efficacy and safety of the intracoronary administration of adrenalin, verapamil, as well as their combination compared to standard treatment in patients with STEMI and refractory coronary no-reflow despite conventional treatment during percutaneous coronary intervention (PPCI)

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PPCI) is the preferred reperfusion strategy for treating acute ST-segment elevation myocardial infarction (STEMI). The main goals are to restore epicardial infarct-related artery patency and to achieve microvascular reperfusion as early as possible. No-reflow is the term used to describe inadequate myocardial perfusion of a given coronary segment without angiographic evidence of persistent mechanical obstruction of epicardial vessels and it refers to the high resistance of microvascular blood flow encountered during opening of the infarct-related coronary artery. Despite optimal evidence-based PPCI, myocardial no-reflow can still occur, negating many of the benefits of restoring culprit vessel patency, and is associated with a worse in-hospital and long-term prognosis.

According to clinical guidelines, nitrates, adenosine, platelet IIb / IIIa receptor inhibitors and thrombus extraction can be used to prevent and treat this complication.These methods have demonstrated the ability to improve coronary blood flow in experiment and small clinical trials, however, limiting the zone of myocardial necrosis and improving disease outcomes have not been achieved.

The search for new methods of influencing the pathogenetic links of this complication is urgent. One of the main potentially reversible factors in the pathogenesis of the no-reflow phenomenon, along with microvascular obstruction, is microvascular arteriolar spasm. Thus, this problem of emergency cardiology remains relevant and requires further research, new methods of prevention and treatment.

Aside from exerting beta-1 agonist properties at higher doses and increasing the inotropic and chronotropic stimulation of the myocardium, epinephrine may, at lower doses, exert potent beta receptor agonist properties that mediate coronary vasodilatation. Another drug with a pronounced coronary vasodilation effect is verapamil.

Based on the pharmacodynamic effects of epinephrine and verapamil, it is expected to increase the vasodilating effect when they are used together, due to the additive type of synergistic interaction, which will improve coronary microcirculation after PCI in patients with acute myocardial infarction and refractory no-reflow phenomenon.

Currently, in clinical practice, there is a possibility of very sensitive diagnosis of microvascular obstruction (MVO) using magnetic resonance imaging (MRI), as well as the area of the coronary reserve according to dynamic perfusion scintigraphy of the myocardium. It is advisable to evaluate the effectiveness of treatment of the no-reflow phenomenon using these methods.

The trial aims to estimate the efficacy and safety of the administration of intracoronary epinephrine, verapamil, as well as their combination versus to standard treatment in patients with STEMI and refractory coronary no-reflow despite conventional treatments during PPCI.

ELIGIBILITY:
Inclusion Criteria:

* patients with ST-elevation myocardial infarction
* Infarct-related artery TIMI flow grade 0-2 during the interventional procedure after the initial opening of the vessel.
* Written the informed consent to participate in research

Exclusion Criteria:

* Unable to undergo or contra-indications for MRI or SPECT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | month 1
  Mortality rate (percent)
New onset or worsening acute heart failure | month 1
  The rate (percent) of patients experiencing new onset or worsening acute heart failure. Congestion characterized by dyspnea, edema, rales, jugular venous distention and need to increase diuretic doses is a hallmark of acute heart failure prompting hospitalization

SECONDARY OUTCOMES:
Thrombolysis in myocardial infarction (TIMI) 3 | hour 1
  The rate of patients (percent) who achieved TIMI 3 coronary blood flow after percutaneous coronary intervention
Change in systolic/diastolic blood pressure | minute 3
  Change in systolic/diastolic blood pressure values (mmHg) before and after intracoronary verapamil/epinephrine
ST segment resolution | hour 72
  Degree of ST segment resolution on ECG (mm)
Troponin I release | hour 72
  Concentration of troponin I (ng/mL)
LV EF | day 10
  Left ventricular ejection fraction (LV EF) (percent)
Myocardial injury | day 2
  Total volume (mL) of microvascular obstruction, myocardial necrosis, edema, and hemorrhagic impregnation according to MRI data
SPECT-based coronary reserve | day 7
  Coronary reserve will be measured by cardiac single photon emission computed tomography (SPECT) with technetium-99m-labeled methoxy-isobutyl isonitrile (99mТсMIBI) at rest and during pharmacological stress-test (counts)
Change in heart rate values | minute 3
  Change in heart rate values (beat per minute) before and after intracoronary verapamil/epinephrine
LV EDV | 10 days
  Left ventricular end-diastolic volume (LV EDV) (mL)
LV ESV | day 10
  Left ventricular end-systolic volume (LV ESV) (mL)
LV WMSI | day 10
  Left ventricular wall motion score index (LV WMSI) (conventional units)
Arrhythmias | minute 5
  Frequency of arrhythmias (atrial fibrillation, atrial flutterу, supraventricular tachycardia, premature ventricular contractions, ventricular tachycardia, conduction disorders and other heart rhythm disorders) after intracoronary administration verapamil and/or epinephrine

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav V Ryabov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk NRMC, Tomsk, Tomsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dil S, Ryabov V, Maslov L, Mochula O, Mochula A, Kercheva M, Zavadovsky K, Vyshlov E. Assessing coronary microvascular dysfunction in refractory no-reflow: Insights from dynamic myocardial perfusion scintigraphy and cardiac MRI. Microvasc Res. 2025 Nov;162:104862. doi: 10.1016/j.mvr.2025.104862. Epub 2025 Aug 20. PMID 40846132